CLINICAL TRIAL: NCT00449800
Title: Pharmacokinetics Variability of Ceftriaxone in Septic ICU Patients
Brief Title: Pharmacokinetic of Ceftriaxone in Septic ICU Patients
Acronym: PORTHOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Pour La Promotion A Tours De La Reanimation Medicale (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APTRM 2006-02
Record Dates: First submitted 2007-03-14; First posted 2007-03-21 (Estimated); Last update posted 2007-03-21 (Estimated); Status verified 2007-03

CONDITIONS: Sepsis; Severe Sepsis; Septic Shock
Keywords: Sepsis; Ceftriaxone; Pharmacokinetic; Intensive care unit
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ceftriaxone

SUMMARY:
Ceftriaxone pharmacokinetics variability in intensive care unit septic patients

In intensive care units, drug dosage is often based on study made on healthy volunteers or on less severe patients.

However, pharmacokinetic alterations have been described for some drugs used in intensive care units.

These alterations, consequences of alteration of volume of distribution, of protein concentrations, of impaired hepatic and renal functions can result in accumulation with toxicity or " under dosage " with inefficacity.

Ceftriaxone is an antibiotic often prescribed in intensive care unit. However, despite this large utilisation, very few data is available on the pharmacokinetic in intensive care unit, and optimal dosage is not known.

Our objective is to develop a population pharmacokinetics model of ceftriaxone in intensive care unit patients with sepsis, severe sepsis and septic shock and to identify the " data " explaining interindividual variability of each pharmacokinetics parameter.

DETAILED DESCRIPTION:
This is a one centre population pharmacokinetics non interventional study. One group of 50 patients allows the development of the model and a second group of 20 patients will be used for the validation of the model.

Septic patients treated with ceftriaxone according to standard procedure of our ICU could be included before the second administration of the drug. In the development group, patients will underwent five determination of serum concentration of ceftriaxone during the 24 hours following the second administration. The timing of samples will be randomised in three groups. A second phase of sampling will take place during the fifth day of ceftriaxone therapy for sepsis and severe sepsis patients and after 48 hours catecholamine- free for septic shock patients.

For the validation group, ten samples will be obtained at the same periods. This study will not induce any change in the care of patients.

Samples will be centrifugated immediately after collection and conserved at - 20 °C.

Ceftriaxone will be assayed in the department of pharmacology, university of Marseille France, usig HPLC method.

Pharmacokinetic analysis will used NONlinear Mixed Effects Modelling logiciel

ELIGIBILITY:
Inclusion Criteria:

* Eighteen-year or more
* sepsis, severe sepsis or septic shock (according to Bone's criteria)
* admission to intensive care unit
* informed consent obtained
* affiliation to medicare

Exclusion Criteria:

* Previous haemodialysis
* hemopathy
* known allergy to cephalosporin
* patients whose death is considered imminent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2006-07; Study Completion 2007-03 (Estimated)

PRIMARY OUTCOMES:
serum drug concentration
pharmacokinetics parameter (plasmatic half-life, clearance, ...)
ratio of serum drug concentration on MCI

CONTACTS AND LOCATIONS:
Overall Officials: DENIS GAROT, MD, Principal Investigator — CHRU TOURS
Locations (1):
- Cenrte Hospitalier Régional Universitaire, Tours, France

REFERENCES:
- [Derived] Garot D, Respaud R, Lanotte P, Simon N, Mercier E, Ehrmann S, Perrotin D, Dequin PF, Le Guellec C. Population pharmacokinetics of ceftriaxone in critically ill septic patients: a reappraisal. Br J Clin Pharmacol. 2011 Nov;72(5):758-67. doi: 10.1111/j.1365-2125.2011.04005.x. PMID 21545483